CLINICAL TRIAL: NCT05618977
Title: The Effect of Dramatization Simulation on Nursing Students' Ethical Attitudes: A Mixed Method Research
Brief Title: The Effect of Dramatization Simulation on Nursing Students' Ethical Attitudes
Acronym: Ethical
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Yadigar Ordu, Lecturer Dr., Çankırı Karatekin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: CankırıKU.
Record Dates: First submitted 2022-10-31; First posted 2022-11-16 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: ETIC

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): In-class case studies will be conducted.
  Interventions: Behavioral: In-class case studies
- Experimental (Experimental): Case studies will be done in the form of dramatization simulation.
  Interventions: Behavioral: Dramatization simulation

INTERVENTIONS:
Behavioral: Dramatization simulation — Ethical attitudes of nursing students will be evaluated with dramatization simulation application.
  Arms: Experimental
Behavioral: In-class case studies — In-class case studies will be conducted with the control group students.
  Arms: Control

SUMMARY:
Nursing students face many ethical problems in their clinical practice. It is very likely that they will encounter ethical problems after graduation. For this reason, students should be given an ethical attitude before graduating. It is very difficult to gain an ethical attitude. Ethical issues, on the other hand, are very difficult to gain as they are a limited concept. Therefore, different methods should be used in teaching. Dramatization simulation is one of the teaching methods used recently. It is especially effective in making abstract concepts that are difficult to understand concrete. It is thought that students participating in a dramatized simulation will be effective in gaining ethical attitudes by recognizing ethical problems more easily. This research will be carried out to determine the effect of dramatization simulation on the ethical attitudes of nursing students.

DETAILED DESCRIPTION:
The effect of dramatization simulation on the ethical attitudes of nursing students will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Students who agreed to participate in the study

Exclusion Criteria:

* Not participating in dramatization simulation applications,
* Not participating in classroom ethical case studies

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Ethical attitude | Four weeks
  Ethical attitudes of nursing students will be determined by using the ethical principles attitude scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Cankiri Karatekin University, Çankırı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No